CLINICAL TRIAL: NCT05307068
Title: Investigation of the Relationships and Clinical Parameters Between IL-10, IL-12 and IL-18 Levels in the Gingival Crevicular Fluid of Individuals With Grade B-C Stage III-IV Periodontitis
Brief Title: IL-10, IL-12 and IL-18 Levels in the Gingival Crevicular Fluid of Patients With Periodontitis and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Elif ilke Cebesoy, PhD student, Istanbul University
Other Study IDs: 679625
Record Dates: First submitted 2022-01-24; First posted 2022-04-01 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis
Keywords: periodontitis; healthy gingiva; grade b; grade c; stage III; stage IV
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Biospecimen Retention: Samples Without DNA — Gingival Crevicular Fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grade B-C stage III-IV periodontitis group: Grade B: Moderate Moderate bone loss is observed compared to biofilm and % Root Bone Loss/age 0.25 to 1.0 is determined as grade B.
  Stage III: Severe Consisted of individuals with interdental AL ≥5 mm, radiographic bone lose extending to middle or apical third of the root, PD≥6 mm and tooth loss due to periodontitis of ≤4.
  Grade C: Rapid Rapid bone loss is observed compared to biofilm and % Root Bone Loss/age >1.0 is determined as grade C.
  Stage IV:Advanced Consisted of individuals with interdental AL ≥5 mm, radiographic bone lose extending to middle or apical third of the root, PD≥6 mm and tooth loss due to periodontitis of ≥5. Need for complex rehabilition due to: Masticatory dysfunction, Secondary occlusal trauma(tooth mobility degree ≥2) Severe ridge defect,Bite collapse, drifting, flaring. Less than 20 remaining teeth (10 opposing pairs)
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis ( periodontitis, healthy)
- Healthy control group: Consisted of individuals with clinically healthy gingiva on an intact periodontium who had a BOP score less than 10% and PD≤3mm, showed no attachment loss or radiographic bone loss.
  Interventions: Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis ( periodontitis, healthy)

INTERVENTIONS:
Other: No intervention was applied to the groups the samples will be collected in terms of the diagnosis ( periodontitis, healthy) — No intervention was applied to the groups the samples will be collected in terms of the diagnosis (periodontitis, healthy)

SUMMARY:
Periodontitis is a multifactorial chronic inflammatory disease characterized by the destruction of the tissues supporting the tooth. The incidence and rate of progression of periodontal destruction involves a complex interaction between periodontopathic bacteria and immune system cells. The complex cytokine network that mediates the immune response includes pro-inflammatory cytokines, anti-inflammatory cytokines, and specific cytokine receptors. Cytokines act as messengers to initiate, mediate, and control immune and inflammatory responses. It is known that the interaction of pro- and anti-inflammatory cytokines plays a very important role in the progression of periodontitis .

The immune response to infection is regulated by the balance between T helper (Th)1 and Th2-type cytokines. Since Th1, Th2, and monocyte-derived cytokines in gingival tissues and gingival crevicular fluid (GCF) play a role in periodontal inflammation, even a minimal imbalance in cytokine production may affect the induction of bone and collagen resorption in periodontal disease. For this reason, cytokines in inflamed periodontal tissues, which are the focus of many studies, are of great importance in the progression of periodontal disease.

In this study, our aim is to evaluate the local cytokine response in relation to the clinical periodontal status by determining the IL-10, IL-12 and IL-18 concentrations in the gingival crevicular fluid of individuals with grade B-C stage III-IV periodontitis according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions. In this way, besides clinical and radiographic determinations in the diagnosis of periodontal disease, IL-10, IL-12 and IL-18 are measured to evaluate whether these markers have an effect on the diagnosis of the disease.

DETAILED DESCRIPTION:
Interleukin-10 (IL-10) is one of the most potent anti-inflammatory cytokines, as it induces T cell anergy (non-responsiveness to an antigen) and reduces the production of some pro-inflammatory cytokines. Altered expression of IL-10, however, genetic predisposition and the presence of specific periodontal bacteria may contribute to the disruption of the Th1/Th2 balance and the development of aggressive periodontitis.

Interleukin-12 (IL-12) is a heterodimer comprised of p35 and p40 subunits, which form the bioactive IL-12 (p70). IL-12 is an essential mediator of the early innate immune response and a key inducer of cellular immunity. Its most important task is to stimulate T cells and interferon-γ (IFN-γ) production by natural killer cells, thereby promoting Th1 responses. The importance of IL-12 is not limited to initiating an immune response, it may contribute to the maintenance of immunity. Because in the absence of IL-12, Th1 responses are rapidly lost.

Interleukin-18 (IL-18) is a pro-inflammatory cytokine belonging to the IL-1 cytokine family. This cytokine was originally identified as a natural killer and a cytokine that induces IFN-γ produced by T cells. IL-18 acts synergistically with IL-12 to support IFN-γ production and Th1 cell growth, but does not depend on IL-12 for its activity.

When this information is brought together, the evaluation of the effects of IL-10, IL-12 and IL-18 concentrations in the gingival crevicular fluid on periodontal disease together with clinical parameters has been the point of our study.

It is planned to include 30 periodontally healthy individuals with grade B-C stage III-IV periodontitis according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions, who applied to Istanbul University Faculty of Dentistry Periodontology Department, after clinical and radiographic evaluations. All individuals to be included will be informed about the purpose and method of the study and their consent will be obtained.

Before the study, it will be ensured that the oral condition of the individual is not caused by any other factor (unknown systemic disease, blood disease, etc.). The individuals included in the study; systemic and oral anamnesis, smoking status, systemic disease status will be recorded and the following clinical measurements will be made.

Gingival crevicular fluid (GCF) samples will be taken from individuals suitable for the study model, and periodontal indices will be recorded. The levels of IL-10, IL-12 and IL-18 will be determined in the GCF samples taken. The researcher will not include individuals who have been included in other studies that have passed or will be approved by the ethics committee, and will not include individuals who will be included in this study, undertakes not to include it in its work.

Clinical measurements include Plaque Index (PI), Gingival Index (GI), Bleeding on Probing (BOP), Probing Depth (PD), Free Gingival Margin (FGM), Clinical Attachment Level Measurement (CAL), Mobility parameters. The measurements were made by the same researcher from six different points of all teeth: mesio-buccal, mid-buccal, disto-buccal, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal. It will be measured and recorded by a single person with the Williams (Hu-Friedy, USA) type periodontal probe. These measurements are non-invasive and will enable us to determine the periodontal status. After the clinical examination and measurements of the patients who met the inclusion criteria and signed the voluntary consent form, the gingival crevicular fluid samples to be taken from the patients will be analyzed and the results will be evaluated. Samples will be isolated from the gingival groove with the aid of absorbent paper strips (Periopaper®, Proflow Inc., Amitiyville, NY, USA) and biochemical analyzes will be made in the samples obtained by ELISA method in accordance with the protocols included in the kit. Biochemical analyzes will be carried out at Istanbul University, Istanbul Faculty of Medicine, Department of Medical Biochemistry.

The clinical evaluation methods planned to be applied in the study are listed below:

1. Plaque Index
2. Probing Depth
3. Bleeding on Probing
4. Clinical Attachment Level Measurement
5. Free Gingival Margin
6. Gingival Index
7. Mobility Samples of paper strips (Periopaper®, Proflow Inc., Amitiyville, NY, USA) placed in the gingival groove will be placed in eppendorf tubes for laboratory examination in the session 1 week after the exact periodontal status is determined by periodontal measurements. Samples will be taken from areas with the deepest probable pocket depth. While obtaining gingival crevicular fluid samples, the area will be isolated with cotton pads and the microbial dental plaque on the tooth will be removed with cotton pellets, and then a short-term drying process will be done with air freshener from a 20 cm distance at a right angle. Then, standard absorbent 2x8 mm paper strips will be placed from the approximal regions to the entrance of the groove with slight resistance and after waiting for 30 seconds, each paper strip will be placed in an eppendorf tube and stored at -80°C. (New Brunswick Scientific Ultra Low Temperature Freezer). Samples will be taken from 6 teeth in each patient.

In case of bleeding from the gingival groove during sample collection, the sample will not be taken from that area.

GCF samples taken and stored at -80°C will be analyzed at Istanbul University, Istanbul Medical Faculty, Department of Medical Biochemistry. IL-10, IL-12 and IL-18 levels of GCF samples will be determined by ELISA method.

In the light of the data, the clinical conditions and biochemical analyzes of the patients will be compared and the relationship between them will be examined.

According to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions, an average of 11 units difference between the results obtained from interleukin biomarkers in the group of individuals with grade B-C stage III-IV periodontitis and healthy individuals, and a minimal sample to find the estimated 15-unit standard deviation significant size (assuming Type I error 5%, Type II error 20% assuming Power 0.80): 30 people for each group. Considering the wrong samples, 30+30 people will be taken into each group (30 healthy controls, 30 Periodontitis cases) Our study will be carried out on systemically healthy patients aged 18-65 years who were diagnosed with Grade B-C stage III-IV periodontitis according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions in the Periodontology Clinic of Istanbul University Faculty of Dentistry.

After the clinical examination and measurements of the patients who met the inclusion criteria and signed the voluntary consent form, the gingival crevicular fluid samples taken from the patients will be analyzed and the results will be evaluated. The samples will be isolated from the gingival crevicular with the help of the absorbent periopaper and biochemically analyzed with ELISA kits.

Periodontitis group:

* 18-65 years old
* Not having any systemic disease (diseases that do not affect the periodontal status)
* Non-smoker
* Have not received antibiotic treatment and/or used immunosuppressant medication in the last 6 months
* Have not received any periodontal treatment in the last 6 months
* No pregnancy and lactation
* Not using any medication regularly
* Having at least 20 teeth
* Grade B-C stage III-IV periodontal disease according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions

Healthy Group:

In patients who applied to Istanbul University Faculty of Dentistry, Department of Periodontology, periodontally healthy individuals who do not meet the above disease criteria, who do not have a history of periodontitis in any way, will be included in the study. Consisted of individuals with clinically healthy gingiva on an intact periodontium who had a BOP score less than 10% and PD≤3mm, showed no attachment loss or radiographic bone loss.

ELIGIBILITY:
Inclusion Criteria for grade B-C stage III-IV periodontitis group:

* 18-65 years old
* Not having any systemic disease (diseases that do not affect the periodontal status)
* Non-smoker
* Have not received antibiotic treatment and/or used immunosuppressant medication in the last 6 months
* Have not received any periodontal treatment in the last 6 months
* No pregnancy and lactation
* Not using any medication regularly
* Having at least 20 teeth
* Grade B-C stage III-IV periodontal disease according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions

Inclusion Criteria for periodontal healthy group:

•In patients who applied to Istanbul University Faculty of Dentistry, Department of Periodontology, periodontally healthy individuals who do not meet the above disease criteria, who do not have a history of periodontitis in any way, will be included in the study. Consisted of individuals with clinically healthy gingiva on an intact periodontium who had a BOP score less than 10% and PD≤3mm, showed no attachment loss or radiographic bone loss.

Exclusion Criteria:

* Those with systemic modifying disease affecting periodontal status
* Smoker
* Have received antibiotic therapy or immunosuppressive therapy in the last 6 months
* Previously received periodontal treatment in the last 6 months
* Pregnancy and breastfeeding status
* Regular use of drugs that will affect systemic health

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In our study individuals who have Grade B-C stage III-IV periodontal disease according to the 2017 Classification of Periodontal and Peri-implant Diseases and Conditions and individuals who have healthy gingiva will be selected
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement of GCF samples | GCF samples were collected after first week of clinical periodontal measurement. GCF was obtained using paper strips from the deepest gingival groove
  Measurement of IL-10, IL-12, IL-18 levels in GCF with grade B-C stage III-IV periodontitis individuals

SECONDARY OUTCOMES:
Measurement of GCF samples | GCF samples were collected after first week of clinical periodontal measurement. GCF was obtained using paper strips from the deepest gingival groove
  Measurement of IL-10, IL-12, IL-18 levels in GCF with periodontal healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Emine Çifcibaşı, Assoc. Prof., Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only clinical istatical analyses and GCF samples analyses will be shared

REFERENCES:
- [Result] Geng Y, Li L, Wang X, He F, Zhou Y, Yang M, Xu Y. Interleukin-10 polymorphisms affect the key periodontal pathogens in Chinese periodontitis patients. Sci Rep. 2018 Jun 13;8(1):9068. doi: 10.1038/s41598-018-26236-4. PMID 29899423
- [Result] Borilova Linhartova P, Danek Z, Deissova T, Hromcik F, Lipovy B, Szaraz D, Janos J, Fassmann A, Bartova J, Drizhal I, Izakovicova Holla L. Interleukin Gene Variability and Periodontal Bacteria in Patients with Generalized Aggressive Form of Periodontitis. Int J Mol Sci. 2020 Jul 2;21(13):4728. doi: 10.3390/ijms21134728. PMID 32630798
- [Result] Orozco A, Gemmell E, Bickel M, Seymour GJ. Interleukin-1beta, interleukin-12 and interleukin-18 levels in gingival fluid and serum of patients with gingivitis and periodontitis. Oral Microbiol Immunol. 2006 Aug;21(4):256-60. doi: 10.1111/j.1399-302X.2006.00292.x. PMID 16842511
- [Result] Pai B S, Pradeep AR. Correlations between Interleukin-33 and -1alpha Levels in Gingival Crevicular Fluid and Plasma in Patients with Chronic or Aggressive Periodontitis and Disease-free Subjects. Bull Tokyo Dent Coll. 2019 Dec 10;60(4):279-289. doi: 10.2209/tdcpublication.2019-0002. Epub 2019 Nov 22. PMID 31761881
- [Result] Park AY, Scott P. Il-12: keeping cell-mediated immunity alive. Scand J Immunol. 2001 Jun;53(6):529-32. doi: 10.1046/j.1365-3083.2001.00917.x. PMID 11422900
- [Result] Clarke IJ, Tilbrook AJ, Galloway DB, Earl CR, Findlay JK, de Kretser DM. Inhibin in rams. J Reprod Fertil Suppl. 1991;43:163-70. No abstract available. PMID 1843338